CLINICAL TRIAL: NCT03263988
Title: A Novel Method of Hemodynamic Monitoring by Piezocapacitative Interlayer Sensor Technology - A Pilot Study
Brief Title: HD Sense Pilot Study - A Novel Method of Hemodynamic Monitoring
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Prof. Dr. med./ Deputy head of department, Charite University, Berlin, Germany
Other Study IDs: HD Sense
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hemodynamic Instability
Keywords: pulse contour analysis; capton; intraoperative monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PIEZO-Group: All patients in this study receive IBP by PICCO and piezocapacitative-interlayer-technology measurement.
  Interventions: Device: ConCardiac

INTERVENTIONS:
Device: ConCardiac — All patients receive a piezocapacitative-interlayer-technology hemodynamic measurement by ConCardiac device (SectorCon GmbH, Berlin, Germany).

SUMMARY:
Measurement of arterial blood pressure is a basic monitoring in the perioperative setting. It is a standard monitoring to assure an adequate cerebral perfusion pressure and is a basic parameter of hemodynamic optimization. Until now standard methods for blood pressure measurement are non-invasive interval monitoring by arm cuff (Riva-Rocci) or direct, continuous and invasive by inserting an intraarterial catheter. This observational study will show, that a new non-invasive piezocapacitative-interlayer technology will make continuous blood pressure monitoring and non-invasive pulse contour analysis available.

DETAILED DESCRIPTION:
Measurement of arterial blood pressure is a basic monitoring in the perioperative setting. It is a standard monitoring to assure an adequate cerebral perfusion pressure and is a basic parameter of hemodynamic optimization. Until now standard methods for blood pressure measurement are non-invasive interval monitoring by arm cuff (Riva-Rocci) or direct, continuous and invasive by inserting an intraarterial catheter. This observational study will show, that a new non-invasive piezocapacitative-interlayer technology will make continuous blood pressure monitoring and non-invasive pulse contour analysis available. For this reason all patients will get a basic monitoring (NIBP, ECG, SpO2)

ELIGIBILITY:
Inclusion Criteria:

* elective surgery and general anesthesia
* age >/= 18 years
* any surgery in ENT/trauma/gynecology/visceral surgery/thoracic surgery/urology/neuro surgery/cardio surgery (N=10)
* cardio surgery (N=10)
* Transcatheter Aortic Valve Implantation (N=20)
* cystectomy (N=10)
* neurosurgery with an expected postoperative ICU stay >/= 20 hours (N=10)

Exclusion Criteria:

* pregnant or breastfeeding patients
* emergency surgery
* participation in a clinical interventional study
* BMI >35 kg/m²
* impossibility to place the ConCardiac interlayer
* difference of blood pressure of right and left arm > 12 mmHg
* pAVK Fontaine IV
* arrythmia absoluta
* vitium cordis >/=3
* ejection fraction <35%
* TAPSE </=16mm
* need of IABP

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years or older voluntary patients undergoing elective surgery at Charité - Universitätsmedizin Berlin Campus Charite Mitte
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PPV | Duration of surgery and perioperative care (an average of 24 hours)
  Percentual error of PPV < 30% for ConCardiac between ConCardiac and PICCO

SECONDARY OUTCOMES:
Duration of surgery | Duration of surgery (an average of 4 hours)
Duration of anesthesia | Duration of surgery (an average of 4 hours)
intraoperative blood loss | Duration of surgery and perioperative care (an average of 24 hours)
Duration of mechanical ventilation | Duration of surgery (an average of 4 hours)
Duration of renal replacement therapy | perioperative (an average of 10 days)
Length of hospital stay | perioperative (an average of 10 days)
Blood products and volume needed perioperative | perioperative (an average of 10 days)
ICU scores (TISS) | perioperative (an average of 10 days)
ICU scores (SOFA) | perioperative (an average of 10 days)
ICU scores (SAPS) | perioperative (an average of 10 days)
Incidence of organ failure or complications | perioperative (an average of 10 days)
Vital signs of patients/blood pressure | perioperative (an average of 10 days)
  RR
Vital signs of patients/heart frequency | perioperative (an average of 10 days)
  HF
Vital signs of patients/Cardiac index | perioperative (an average of 10 days)
  CI
Vital signs of patients/stroke volume | perioperative (an average of 10 days)
  SV
Vital signs of patients/pulse pressure variation | perioperative (an average of 10 days)
  PPV
Vital signs of patients/systemic vascular resistance index | perioperative (an average of 10 days)
  SVRI
Vital signs of patients/intrathoracic blood volume index | perioperative (an average of 10 days)
  ITBV/I
Vital signs of patients/extra vascular lung water index | perioperative (an average of 10 days)
  ELWI
Vital signs of patients/global enddiastolic volume index | perioperative (an average of 10 days)
  GEDI
Vital signs of patients/Ventilator settings | perioperative (an average of 10 days)
  Ventilator settings
Vital signs of patients/blood gases | perioperative (an average of 10 days)
  BGA
Vital signs of patients/creatinine | perioperative (an average of 10 days)
  Creatinine
Vital signs of patients/central venous oxygen saturation | perioperative (an average of 10 days)
  ScvO2
Vital signs of patients/central venous pressure | perioperative (an average of 10 days)
  CVP
Vital signs of patients/diuresis | perioperative (an average of 10 days)
  Diuresis

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Treskatsch, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin Campus Charité Mitte, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807
- [Background] Scheer B, Perel A, Pfeiffer UJ. Clinical review: complications and risk factors of peripheral arterial catheters used for haemodynamic monitoring in anaesthesia and intensive care medicine. Crit Care. 2002 Jun;6(3):199-204. doi: 10.1186/cc1489. Epub 2002 Apr 18. PMID 12133178
- [Background] Scheeren TW, Wiesenack C, Gerlach H, Marx G. Goal-directed intraoperative fluid therapy guided by stroke volume and its variation in high-risk surgical patients: a prospective randomized multicentre study. J Clin Monit Comput. 2013 Jun;27(3):225-33. doi: 10.1007/s10877-013-9461-6. Epub 2013 Apr 5. PMID 23558909
- [Background] Auler JO Jr, Galas F, Hajjar L, Santos L, Carvalho T, Michard F. Online monitoring of pulse pressure variation to guide fluid therapy after cardiac surgery. Anesth Analg. 2008 Apr;106(4):1201-6, table of contents. doi: 10.1213/01.ane.0000287664.03547.c6. PMID 18349193
- [Background] Dalfino L, Giglio MT, Puntillo F, Marucci M, Brienza N. Haemodynamic goal-directed therapy and postoperative infections: earlier is better. A systematic review and meta-analysis. Crit Care. 2011 Jun 24;15(3):R154. doi: 10.1186/cc10284. PMID 21702945
- [Background] Sun Y, Lacour SP, Brooks RA, Rushton N, Fawcett J, Cameron RE. Assessment of the biocompatibility of photosensitive polyimide for implantable medical device use. J Biomed Mater Res A. 2009 Sep 1;90(3):648-55. doi: 10.1002/jbm.a.32125. PMID 18563817